CLINICAL TRIAL: NCT06984081
Title: CAPA In-vitro Oocyte Maturation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Pui Wah Jacqueline, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CREC.2025.238
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Infertility, Female
Keywords: In Vitro Oocyte Maturation Techniques
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPA-IVM (Experimental): In CAPA-IVM, the oocyte is treated and matured outside the woman's body, while in classical IVF, the patient is treated. As a consequence, patients undergoing CAPA-IVM are not confronted with the typical risks and burden of systemic ovarian stimulation.
  Interventions: Procedure: CAPA IVM

INTERVENTIONS:
Procedure: CAPA IVM — In CAPA-IVM, the oocyte is treated and matured outside the woman's body, while in classical IVF, the patient is treated. As a consequence, patients undergoing CAPA-IVM are not confronted with the typical risks and burden of systemic ovarian stimulation.

SUMMARY:
In vitro oocyte maturation (IVM) is a mild-approach assisted reproductive technology (ART). Because of its simplicity, the more favorable financial implications (reduced cost) for patients, and the lower health risk profile of IVM compared to controlled ovarian stimulation (COS) in polycystic ovary syndrome (PCOS) patients, the use of IVM in selected patients may gain increasing interest. Besides its application in patients with polycystic ovaries, IVM technology may have a role in fertility preservation, where young girls and adult women are facing infertility due to gonadotoxic chemotherapeutic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 0-50 years old
* Patients seek fertility preservation services
* Patients seek oocyte retrieval services

Exclusion Criteria:

-Patients unable to provide consent/assent (i.e. significant psychiatric problems/cognitive delay)

Ages: 0 Months to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2030-05-31 (Estimated); Study Completion 2032-05-31 (Estimated)

PRIMARY OUTCOMES:
No. of mature oocytes | 1 week
  Number of mature oocytes after IVM

CONTACTS AND LOCATIONS:
Overall Officials: Pui Wah Jacqueline Chung, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No